CLINICAL TRIAL: NCT04392284
Title: Using the Sequential Multiple Assignment Randomized Trial Experimental Approach to Develop an Adaptive Lifestyle Intervention Program in Family Medicine Clinics
Brief Title: Developing an Adaptive Lifestyle Intervention Program in Family Medicine Clinics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Drew Sayer, Primary Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300005391
Record Dates: First submitted 2020-04-19; First posted 2020-05-18 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Insulin Resistance; Obesity; Diabetes; Hypertension; Dyslipidemias; Metabolic Syndrome
Keywords: insulin resistance
MeSH Terms: conditions — Insulin Resistance; Obesity; Diabetes Mellitus; Hypertension; Dyslipidemias; Metabolic Syndrome

STUDY DESIGN:
Intervention Model Description: Sequential Multiple Assignment Randomized Trial (SMART)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet Counseling (Experimental): Delivery of nutrition counseling intervention to improve diet quality.
  Interventions: Behavioral: Diet Counseling
- Exercise Counseling (Experimental): Delivery of exercise counseling intervention to increase engagement in physical activity..
  Interventions: Behavioral: Exercise Counseling

INTERVENTIONS:
Behavioral: Diet Counseling — Delivery of nutrition counseling intervention to improve diet quality. Suggested energy intake will be prescribed with the intent to maintain energy balance and current body weight. A total of 16 nutrition counseling sessions lasting ~30 minutes will be scheduled with a frequency of 1 session per week for 1 month (5 sessions), 1 session every-other week for months 2-6 (11 sessions). "Responding" participants who have improved their insulin resistance as measured at the 8-week visit will continue receiving this level of nutrition counseling through the end of the study, meeting with the dietitian every other week. Starting at week 9, those identified as "non-responding" participants will be re-randomized to 2nd stage interventions, of either receiving nutrition counseling for weight loss (meeting with the dietitian every other week) or the addition of a prescription for metformin.
  Arms: Diet Counseling
Behavioral: Exercise Counseling — Delivery of exercise counseling intervention to increase engagement in physical activity. The exercise specialist will counsel participants to progressively increase their weekly physical activity. Weight loss is not a primary goal of these exercise counseling sessions. A total of 16 exercise counseling sessions lasting ~30 minutes will be scheduled with a frequency of 1 session per week for 1 month (5 sessions), 1 session every-other week for months 2-6 (11 sessions). "Responding" participants who have improved their insulin resistance as measured at the 8-week visit will continue receiving this level of exercise counseling through the end of the study, meeting with the exercise specialist every other week. Starting at week 9, those identified as "non-responders" will be re-randomized to 2nd stage interventions, of either receiving nutrition counseling for weight loss (meeting with the dietitian every other week) or the addition of a prescription for metformin.
  Arms: Exercise Counseling

SUMMARY:
The purpose of this study is to investigate the feasibility of conducting a multicomponent lifestyle intervention research study within the UAB Family Medicine Clinic at Highlands and to obtain preliminary data on the effectiveness of the adaptive treatment strategies being investigated to produce improvements in insulin resistance. This study is a Sequential Multiple Assignment Randomized Trial (SMART) with initial randomization groups of individualized nutrition counseling vs. individualized exercise counseling. Note that these initial nutrition or exercise interventions are NOT intended to produce significant weight loss. Participants that do not sufficiently improve their insulin resistance score after 8 weeks will be re-randomized to 2nd stage interventions of either receiving dietary counseling for weight loss or receiving a prescription for metformin. We will collect data on the effectiveness of the intervention to improve insulin resistance/metabolic health in the family medicine clinic as well as potential predictors or moderators of treatment success.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Any race or ethnicity
* BMI >27 kg/m2
* Presence of 1 or more mild-to-moderate obesity-associated metabolic complications (i.e., Stage 1 Obesity)
* Prediabetes, type 2 diabetes (see exclusion criteria for additional details), metabolic syndrome, dyslipidemia, hypertension, non-alcoholic fatty liver disease
* Stable medication type and dosage for ≥3 months

Exclusion Criteria:

* If type 2 diabetes,
* Currently prescribed metformin or prescribed within previous 3 months
* HbA1c concentration of >12%
* Using exogenous insulin
* Pregnant or lactating within the past 6 months or trying to become pregnant
* Prescription for weight loss medications within the past 3 months
* Severe obesity-related complications that require immediate and more intensive clinical therapy (e.g., pharmacotherapy and/or bariatric surgery) as determined by study physician and/or referring practitioner at UAB Family Medicine Clinic.
* History of kidney disease that may increase the risk of lactic acidosis with metformin.
* Currently prescribed the following medications that may increase the risk of lactic acidosis with metformin: acetazolamide (Diamox), dichlorphenamide (Keveyis), methazolamide, topiramate (Topamax, in Qsymia), or zonisamide (Zonegran).
* Does not have a life-sustaining medical implant such as a pacemaker.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-03 (Actual)

PRIMARY OUTCOMES:
Rates of recruitment and retention | Baseline
  Number of participants recruited and retained in intervention
Rates of recruitment and retention | Month 2
  Number of participants recruited and retained in intervention
Rates of recruitment and retention | Month 6
  Number of participants recruited and retained in intervention
Family medicine clinician referral rates | Baseline
Family medicine clinician referral rates | Month 2
Family medicine clinician referral rates | Month 6
Number of counseling sessions attended | Month 2
  Attendance to Zoom meetings
Number of counseling sessions attended | Month 6
  Attendance to Zoom meetings
Frequency of metformin adherence (as applicable) | Month 2
  Number of times metformin was taken as prescribed
Frequency of metformin adherence (as applicable) | Month 6
  Number of times metformin was taken as prescribed
Intervention preference | Baseline
  Preference is determined by the Intervention Preference Questionnaire, using a 5-point Likert Scale for preference among study treatment arms. Scale includes options for "strong," "slight," or "no" preference for a given treatment component.
Intervention preference | Month 2
  Preference is determined by the Intervention Preference Questionnaire, using a 5-point Likert Scale for preference among study treatment arms. Scale includes options for "strong," "slight," or "no" preference for a given treatment component.
Intervention preference | Month 6
  Preference is determined by the Intervention Preference Questionnaire, using a 5-point Likert Scale for preference among study treatment arms. Scale includes options for "strong," "slight," or "no" preference for a given treatment component.
Treatment credibility | Baseline
  Assessment of participants' perception of treatment success using the Credibility/Expectancy Questionnaire with a 9-point Likert scale, ranging from "not at all" (1) to "very" (9) for several descriptors (e.g., "useful," "logical.")
Treatment credibility | Month 2
  Assessment of participants' perception of treatment success using the Credibility/Expectancy Questionnaire with a 9-point Likert scale, ranging from "not at all" (1) to "very" (9) for several descriptors (e.g., "useful," "logical.")
Treatment credibility | Month 6
  Assessment of participants' perception of treatment success using the Credibility/Expectancy Questionnaire with a 9-point Likert scale, ranging from "not at all" (1) to "very" (9) for several descriptors (e.g., "useful," "logical.")

SECONDARY OUTCOMES:
Changes in body weight | Baseline to Months 2 and 6
Changes in body composition (fat and lean mass) | Baseline to Months 2 and 6
  Fat mass and lean mass via bioelectrical impedance analysis
Changes in glucose | Baseline to Months 2 and 6
  Serum glucose will be measured in a fasted state
Changes in insulin | Baseline to Months 2 and 6
  Serum insulin will be measured in a fasted state
Changes in glycosylated hemoglobin (hemoglobin A1C) | Baseline to Months 2 and 6
  Percentage (%) glycated hemoglobin as a measure of long-term blood glucose control
Changes in lipids | Baseline to Months 2 and 6
  Fasting serum concentrations of total cholesterol, LDL cholesterol, HDL cholesterol, and triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Drew Sayer, PhD, Principal Investigator — University of Alabama at Birmingham; Tapan Mehta, PhD, Principal Investigator — University of Alabama at Birmingham; Gareth Dutton, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Highlands Family and Community Medicine Clinic, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No